CLINICAL TRIAL: NCT02891785
Title: Evaluation of the Project "Improvement of Nurse-led Self-management Support for Patients With Cancer-related Pain": An Accompanying Cluster Randomized Study With a Stepped Wedge Design
Brief Title: Praxis Evaluation of a Pain Self-management Support Intervention for Oncology Patients: A Stepped Wedge Design Study
Acronym: EvANtiPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other); University of Lausanne (Other)
Responsible Party: Principal Investigator, Antje Koller, PhD, PhD, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: UVienna
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cancer Pain Self-management
MeSH Terms: interventions — Antipain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ANtiPain intervention (Experimental): ANtiPain is a cancer pain self-management support intervention administered by nurses in an intervention session while the patient is still hospitalized and via phone calls after discharge. ANtiPain is based on three key strategies: information, skill building and nurse coaching.
  Interventions: Behavioral: ANtiPain
- standard care (No Intervention): Standard care will be described as part of the study.

INTERVENTIONS:
Behavioral: ANtiPain — After the implementation of ANtiPain, patients will receive cancer pain self-management support by trained staff nurses who follow the ANtiPain protocol. ANtiPain is based on 3 key strategies: Provision of information, skill building and nurse coaching. It consists of an in-hospital one-to-one session before discharge and a telephone follow up according to a clinical algorithm based on pain intensity, patient satisfaction with pain management and patient adherence. Patients will be given a booklet with corresponding info. The implementation process will include training of designated staff nurses, coaching activities based on case discussions on the ward, as well as measures to ensure sustainability of the implementation (e.g., training of ward managers and clinical nurse specialists).
  Arms: ANtiPain intervention

SUMMARY:
Background: Significant barriers to cancer pain management are patient-related. So far, cancer pain self-management support interventions have only been tested in strictly controlled settings of randomized controlled trials (RCT) and thus evidence for comparative effectiveness is lacking.

Methods: This study includes a multicenter cluster RCT with a stepped wedge design and a qualitative substudy. The aim of the study is to evaluate the implementation of ANtiPain in clinical practice. The primary patient-related aim is to improve pain interference with daily activities. Secondary patient-related aims are pain intensity, barriers to pain management, self-efficacy, and quality of life. Secondary organization-related aims are nurse proficiency and satisfaction with cancer pain self-management support, participation rates, and implementation fidelity.

Inclusion and exclusion criteria: On 17 wards in 3 hospitals in Vienna adult oncology patients will be included (n=150 pre-, n=150 post-implementation) if they are admitted to one of the participating wards, have pain ≥3 (0=no pain to 10=worst imaginable pain) or regular pain medication, able to understand German, discharged with pain self-management, and give informed consent. Patients with signs of disorientation that may severely limit pain self-management will be excluded.

Interventions: Pre-implementation, patients receive standard care. Post-implementation, patients receive ANtiPain which is based on 3 key strategies: information, skills building and nurse coaching and consists of in-hospital sessions by staff nurses and follow-up phone calls after discharge. The implementation process will include training of the designated staff nurses, case discussions, as well as measures to ensure sustainability of the implementation (e.g., training of clinical nurse specialists).

Procedures: Wards are randomized according to the stepped wedge plan. Patients will complete questionnaires at admission, and 2, 4 and 8 weeks after discharge. Nurse-level data will be collected before implementation and 1 and 3 months after implementation. Data on ward and hospital level will be collected at the beginning of the study.

Statistical analysis: The statistical analysis will be conducted based on mixed models, with a random intercept for the respective ward and time as a covariate.

Qualitative substudy: The qualitative substudy will comprise interviews with head and intervention nurses about their views of the implementation.

DETAILED DESCRIPTION:
Background Despite highly effective treatment options, adequate pain control is a persistent problem in oncology patients. As cancer treatment is shifted increasingly towards the outpatient setting, patients' self-management is vital for successful pain treatment. ANtiPain (Advanced Nursing Practice cancer pain self-management support) is a cancer pain self-management support intervention for patients with cancer that is already available and tested in a German speaking setting. So far, cancer pain self-management support interventions have only been tested in the rigorously controlled setting of a randomized controlled trial (RCT) and thus evidence for its comparative effectiveness is lacking.

Objective This study is unique in that it aims to evaluate the implementation of the ANtiPain intervention in routine clinical practice in view of its effectiveness for patients and nurses in realistic clinical settings.

Methods Design, setting and sample In the context of routine quality improvement, AntiPain will be implemented on designated wards at three hospitals in Vienna. To evaluate the implementation, an accompanying multicenter cluster randomized trial with a stepped wedge design will be supplemented with embedded qualitative evaluations. The stepped wedge design will involve the sequential rollout of the intervention. The order in which ANtiPain will be implemented on the wards will be determined at random. By the end of the study, all wards will have implemented the intervention.

Patients will be recruited on 17 wards. With an effect size of d=.77 and an expected drop-out rate of 20%, a sample size of 150 patients will be needed before and after implementation to demonstrate a difference at the 5% level with 90% power. With 17 wards and a study duration of 15 months, approximately 1.3 patients will be recruited per month on each of the participating wards.

Objective and specific aims In congruence with the Reach Efficacy Adoption Implementation and Maintenance (RE-AIM) framework, the implementation of ANtiPain will be evaluated on two levels: (i) patient-related outcomes (e.g., pain interference with daily activities, pain intensity, patient related barriers to cancer pain management), and (ii) organization-related outcomes (e.g., nurses' self-rated perceived proficiency with pain management, application fidelity).

The primary aim of this implementation project is to improve patient-related outcomes. The primary patient-related outcome will be pain interference with daily activities. Secondary patient-related outcomes will be pain intensity, patient-related barriers to cancer pain management, pain-related self-efficacy, and quality of life. The secondary aim is to explore the participation rate [Reach], to improve nurse-related outcomes [e.g. proficiency and satisfaction concerning pain self-management support (Adoption and Implementation)], to achieve high implementation fidelity in the clinical setting [Implementation], to evaluate the nursing managers' view on the implementation [Adoption], a crude cost and resource estimation of the implementation [Adoption], to explore how implementation fidelity will develop over time [Maintenance], and to explore the nursing managers views on maintaining the intervention in their organization [Maintenance]).

Implementation of cancer pain self-management support Before the implementation, patients receive standard care without structured cancer pain self-management support. After implementation, patients will receive cancer pain self-management support by trained staff nurses who follow the ANtiPain protocol. ANtiPain is based on three key strategies: Provision of information, skills building and nurse coaching. It consists of an in-hospital baseline one-to-one session before discharge and a telephone follow up according to a structured clinical algorithm that is based on pain intensity, patient satisfaction with pain management and patient adherence. The implementation process will include training of the designated staff nurses, coaching activities based on case discussions on the ward, as well as measures to ensure sustainability of the implementation (e.g., training of ward managers and clinical nurse specialists).

Variables and Measurement Data collection on patient level will include pain interference with daily activities, pain intensity, and analgesic intake from the Brief Pain Inventory. In addition, the self-developed item from a previous study will be used to measure pain-related activity hindrance, by asking patients to rate "The pain hindered me to do things that I wanted to do today" on a 0 (not at all) to 10 (completely) numeric rating scale. Patient-related barriers to cancer pain management will be measured with the German short version of the Barriers Questionnaire II (BQII-G-S); pain-related self-efficacy with the German version of the Pain Self-efficacy Questionnaire (FESS); HRQoL with two items from the EORTC-Quality of Life Questionnaire C30, functional status with the German version of the Eastern Cooperative Oncology Group Performance Status (ECOG-PS); Depression with the Patient Health Questionnaire (PHQ-2); demographic and clinical data will include age, gender, time since first cancer diagnosis, time since first pain onset, circadian rhythm of pain, and analgesic medication, reason for and day of hospitalization as well as the day of discharge. Full patient self-report data collection will include ~80 items. Because patient burden was a substantial issue in our last studies, patients who say that they cannot complete all questionnaires will be offered to complete a short version of the study questionnaires (49 items).

Data collection on nurse level will include 4 questions regarding self-rated proficiency with cancer pain self-management support and satisfaction with pain management on the ward. In addition, demographic data will be obtained (e.g., age, time on ward). Data collection on ward and hospital level will include the medical field, length of stay, and the number of patients (with cancer-related pain). Standard care will be explored by asking nurses about their role in cancer pain self-management support before the implementation.

Qualitative substudy: The qualitative substudy will comprise interviews with head nurses and intervention nurses about their views of the implementation.

Procedures Wards will be randomized according to the stepped wedge plan. Data collection will start January 2016. Eligible patients will be recruited by staff nurses who will be supported by a study assistant. After informed consent patients will be asked to complete questionnaires at admission (TP0), as well as 2 (TP1), 4 (TP2) and 8 weeks (TP3) after discharge. Nurse-level data will be collected one week before implementation (TN0) and 1 (TN1) and 3 months after implementation (TN2). Data on ward and hospital level will be collected by a study assistant at the beginning of the study.

The statistical analysis of the primary outcome (i.e., pain interference with daily activities) will be conducted based on mixed models, with a random intercept for the respective ward and time as a covariate to take potential time trends into account.

Ethical considerations The study will be conducted in accordance with the Declaration of Helsinki. Within the clusters (wards), patients will be provided with tailored oral and written informed consent (i.e., pre- and post-implementation). During the informed consent procedure patients will be informed about the quality improvement project in general. As soon as the intervention has been implemented in routine clinical practice on the respective ward, patients will be offered the intervention. Consequently, the informed consent procedure will not involve consent for the intervention but only for the completion of questionnaires.

ELIGIBILITY:
Wards

Inclusion Criteria:

* ≥20% of oncology patients
* pre-selection by nursing director and clinical nurse specialists
* willing to participate

Patients

Inclusion Criteria:

* admission to one of the participating wards
* cancer-related pain ≥3 on 11-point numeric rating scale within the last week or
* have regular pain medication because of cancer-related pain
* are able to read and write German
* likely to be discharged with pain self-management
* willing to participate

Exclusion Criteria:

* if patients are showing signs of disorientation that may limit their ability to perform pain self-management at home as assessed by staff nurse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
pain interference with daily activities TP1 | Change from Baseline in pain interference with daily activities at 2 weeks after discharge
  7-item scale from Brief pain Inventory
pain interference with daily activities TP2 | Change from Baseline in pain interference with daily activities at 4 weeks after discharge
  7-item scale from Brief pain Inventory

SECONDARY OUTCOMES:
pain intensity TP1 | Change from Baseline in pain intensity at 2 weeks after discharge
  11-point numeric rating scale (0=no pain; 10=worst imaginable pain)
pain intensity TP2 | Change from Baseline in pain intensity at 4 weeks after discharge
  11-point numeric rating scale (0=no pain; 10=worst imaginable pain)
BQII-G TP1 | Change from Baseline in BQII-G scores at 2 weeks after discharge
  patient related barriers to cancer pain management
BQII-G TP2 | Change from Baseline in BQII-G scores at 4 weeks after discharge
  patient related barriers to cancer pain management
Self Efficacy Scale TP1 | Change from Baseline in Self Efficacy Scale scores at 2 weeks after discharge
  pain-related self-efficacy
Self Efficacy Scale TP2 | Change from Baseline in Self Efficacy Scale scores at 4 weeks after discharge
  pain-related self-efficacy
Health-Related Quality of Life TP1 | Change from Baseline in Health-Related Quality of Life scores at 2 weeks after discharge
  2 11-point numeric rating scales
Health-Related Quality of Life TP2 | Change from Baseline in Health-Related Quality of Life scores at 4 weeks after discharge
  2 11-point numeric rating scales
participation rate | count during study
  number of patients who are asked, versus number of participants who agree to participate in the study/in the intervention at study completion
nurse-related outcomes 1 and 3 months after implementation | Change from before implementation of ANtiPain until 1 and 3 months after implementation
  proficiency and satisfaction concerning pain self-management support
pain interference with daily activities TP3 | Change from Baseline in pain interference with daily activities at 8 weeks after discharge
  7-item scale from Brief pain Inventory
pain intensity TP3 | Change from Baseline in pain intensity at 8 weeks after discharge
  11-point numeric rating scale (0=no pain; 10=worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Antje Koller, PhD, Principal Investigator — University of Vienna, Faculty of Social Sciences, Institute of Nursing Science
Locations (3):
- Austria (3):
  - Krankenhaus Hietzing, Vienna
  - Wilhelminenspital, Vienna
  - Vienna General Hospital, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raphaelis S, Frommlet F, Mayer H, Koller A. Implementation of a nurse-led self-management support intervention for patients with cancer-related pain: a cluster randomized phase-IV study with a stepped wedge design (EvANtiPain). BMC Cancer. 2020 Jun 16;20(1):559. doi: 10.1186/s12885-020-06729-0. PMID 32546177